CLINICAL TRIAL: NCT03612687
Title: Use of an Advanced Minimally Invasive Hemodynamic Monitoring for Perioperative Fluid Management in Hepatobiliary and Pancreas Surgery: A Pilot Study
Brief Title: Hemodynamic Monitoring in Hepatopancreaticobiliary (HPB) Surgery
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 03-14-03E
Record Dates: First submitted 2014-05-22; First posted 2018-08-02 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2018-07

CONDITIONS: Cancer
Keywords: Hemodynamic Monitoring; Perioperative Fluid Management; Hepatobiliary and Pancreas Surgery
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (4):
- Laparoscopic Liver Surgery: Laparoscopic Liver Surgical Procedures with minimally invasive hemodynamic monitoring
  Interventions: Device: Minimally invasive hemodynamic monitoring
- Laparoscopic Pancreas Surgery: Laparoscopic Pancreas Surgical Procedures with minimally invasive hemodynamic monitoring
  Interventions: Device: Minimally invasive hemodynamic monitoring
- Open Liver Surgery: Open Liver Surgical Procedures with minimally invasive hemodynamic monitoring
  Interventions: Device: Minimally invasive hemodynamic monitoring
- Open Pancreas Surgery: Open Pancreas Surgical Procedures with minimally invasive hemodynamic monitoring
  Interventions: Device: Minimally invasive hemodynamic monitoring

INTERVENTIONS:
Device: Minimally invasive hemodynamic monitoring — Use of advanced minimally invasive hemodynamic monitoring with PreSep™ Central Venous Oximetry Catheter, Vigileo™ monitor, and FloTrac™ sensor for perioperative fluid management

SUMMARY:
This is a pilot study with the primary objective to validate the use of advanced minimally invasive hemodynamic monitoring with the PreSep™ Central Venous Oximetry Catheter, the Vigileo™ monitor, and FloTrac™ sensor for perioperative fluid management in Hepatobiliary and Pancreas Surgery. All of these devices and monitors are FDA approved devices and routinely used in the perioperative setting for these cases.

DETAILED DESCRIPTION:
Surgical procedures involving the liver and pancreas are complex and involve paying close attention to hemodynamics to keep the patient stable through the duration of the case. Volume overload in liver and pancreas surgery leads to more intraoperative blood loss and rapid volume shifts make the patient unstable and more difficult to manage. Traditional methods of invasive monitoring to determine cardiac output and stroke volume include the placement of a pulmonary artery catheter and an arterial line. With the addition of the FloTrac™ Sensor to the arterial line and the Vigileo™ monitor; a pulmonary artery catheter would be no longer required. The minimally invasive cardiac output monitor connected to the central venous catheter will generate detailed information of cardiac function and fluid status and thereby help monitor and manage the hemodynamics of the patient intraoperatively. The information obtained from the Vigileo™ will be compared to the regular data normally available in patients undergoing hepatobiliary surgery to determine the advantages of using the system to aid in fluid management of the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female patients admitted to Carolinas Medical Center (CMC) with the need for the following surgical procedures: liver resection, distal pancreatectomy and splenectomy, and pancreaticoduodenectomy.

Exclusion Criteria:

1. Indication for emergency surgery, including pancreatic debridement in an acute setting; ruptured hepatic adenomas/hepatocellular carcinomas
2. Suspected inability to comply with trial procedures or understand consent
3. Employee at the investigational center, relative or spouse of the investigators
4. Patients incarcerated at the time of surgery
5. Females who are pregnant or breastfeeding
6. Planned use of Cell Saver during surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The procedures will be divided by organ systems, liver and pancreas, and by method of surgery, laparoscopic versus open. Five patients will be chosen for each group for a total of 20 patients enrolled. The following procedures will be included in the study: liver resection (>2 segments), distal pancreatectomy and splenectomy, and pancreaticoduodenectomy, including robotic procedures.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Incidence of intraoperative complications | Intraoperative period
  Cardiocirculatory, respiratory, neurological, renal, infectious and major bleeding events

SECONDARY OUTCOMES:
Extubation time | up to 48 hours
  Measurement of time to extubation (hours)
Incidence of postoperative blood transfusions | up to 10 days
  Volume of blood transfused following surgical procedure (mL)
Incidence of postoperative complications | up to 10 days
  Rate of pre-specified postoperative complications (number of patients affected)
ICU length of stay | up to 3 days
  Intensive Care Unit (ICU) length of stay (days)
Length of hospital stay | up to 10 days
  Time to discharge from hospital (days)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Swan, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No